CLINICAL TRIAL: NCT02839668
Title: The Impact of Intravenous Anaesthesia on Angiogenesis in Patients With Breast Cancer
Brief Title: The Impact of Intravenous Anaesthesia on Angiogenesis in Patients With Breast Cancer (TIVA/TCI-BC)
Acronym: TIVA/TCI-BC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Collaborators: Prof. Dr. I. Chiricuta Institute of Oncology (Other)
Responsible Party: Principal Investigator, Dr.Draghiciu Elena, Universitary Assistant, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IuliuHatieganu Cluj-Napoca
Record Dates: First submitted 2016-06-18; First posted 2016-07-21 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; angiogenesis; VEGF
MeSH Terms: conditions — Breast Neoplasms | interventions — Lidocaine; Sevoflurane; Propofol; Acetaminophen; Tramadol; Neostigmine; Atropine; Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sevoflurane (Experimental): The patients enrolled in this arm will receive general anesthesia in which the hypnosis will be maintained with Sevoflurane. Postoperative analgesia will be assured by the administration of tramadol and acetaminophen.A 0.05 mg/kg dose of neostigmine will be administered to antagonize the neuromuscular block at the end of surgery.A 0.2 mg/kg dose of atropine will be administered at the end of surgery to attenuate the parasymatomimetic effects of neostigmine.The bispectral index- BIS will be monitored throughout the anesthesia
  Interventions: Drug: Sevoflurane; Drug: Acetaminophen; Drug: Tramadol; Drug: Neostigmine; Drug: Atropine; Device: BIS
- Sevoflurane+Lidocaine (Active Comparator): The patients enrolled in this group will receive general anesthesia in which the hypnosis will be maintained with Sevoflurane. At the induction of anesthesia the patients will receive a bolus of lidocaine 1% 1.5 mg/kg. A continuous infusion of lidocaine 1% of 2 mg/kg/h will be associated throughout the surgical procedure and 1mg/kg/h until 24 h postoperative. Postoperative analgesia will be assured by the administration of tramadol and acetaminophen.A 0.05 mg/kg dose of neostigmine will be administered to antagonize the neuromuscular block at the end of surgery. A 0.2 mg/kg dose of atropine will be administered at the end of surgery to attenuate the parasymatomimetic effects of neostigmine.The bispectral index- BIS will be monitored throughout the anesthesia
  Interventions: Drug: Lidocaine; Drug: Sevoflurane; Drug: Acetaminophen; Drug: Tramadol; Drug: Neostigmine; Drug: Atropine; Device: BIS
- TIVA-TCI (Experimental): The patients enrolled in this group will receive total intravenous anesthesia with propofol using a target controlled infusion technique for the maintenance of hypnosis throughout the surgery. Postoperative analgesia will be assured by the administration of tramadol and acetaminophen.A 0.05 mg/kg dose of neostigmine will be administered to antagonize the neuromuscular block at the end of surgery.A 0.2 mg/kg dose of atropine will be administered at the end of surgery to attenuate the parasymatomimetic effects of neostigmine. The bispectral index- BIS will be monitored throughout the anesthesia.
  Interventions: Drug: TIVA-TCI; Drug: Acetaminophen; Drug: Tramadol; Drug: Neostigmine; Drug: Atropine; Device: BIS
- TIVA-TCI+lidocaine (Active Comparator): The patients enrolled in this group will receive total intravenous anesthesia with propofol using a target controlled infusion technique for the maintenance of hypnosis throughout the surgery. At the induction of anesthesia the patients will receive a bolus of lidocaine 1% 1.5 mg/kg. A continuous infusion of lidocaine 1% of 2 mg/kg/h will be associated throughout the surgical procedure and 1mg/kg/h until 24 h postoperative. Postoperative analgesia will be assured by the administration of tramadol and acetaminophen.A 0.05 mg/kg dose of neostigmine will be administered to antagonize the neuromuscular block at the end of surgery. A 0.2 mg/kg dose of atropine will be administered at the end of surgery to attenuate the parasymatomimetic effects of neostigmine.The bispectral index- BIS will be monitored throughout the anesthesia.
  Interventions: Drug: Lidocaine; Drug: TIVA-TCI; Drug: Acetaminophen; Drug: Tramadol; Drug: Neostigmine; Drug: Atropine; Device: BIS

INTERVENTIONS:
Drug: Lidocaine — Continuous infusion of lidocaine
  Other Names: lidocaine 1%, lignocaine
  Arms: Sevoflurane+Lidocaine; TIVA-TCI+lidocaine
Drug: Sevoflurane — maintenance of hypnosis during anaesthesia with sevoflurane
  Arms: Sevoflurane; Sevoflurane+Lidocaine
Drug: TIVA-TCI — maintenance of hypnosis during anaesthesia with sevoflurane
  Other Names: Diprivan
  Arms: TIVA-TCI; TIVA-TCI+lidocaine
Drug: Acetaminophen — administration of 1 g acetaminophen for postoperative analgesia
  Other Names: paracetamol
Drug: Tramadol — administration of tramadol for postoperative analgesia
  Other Names: Tramal
Drug: Neostigmine — A 0.05 mg/kg dose of neostigmine will be administered to antagonize the neuromuscular block at the end of surgery.
  Other Names: Prostigmin, vagostigmin
Drug: Atropine — A 0.2 mg/kg dose of atropine will be administered at the end of surgery to attenuate the parasymatomimetic effects of neostigmine
  Other Names: atropine sulfate
Device: BIS — For the groups receveing TIVA-TCI anesthesia the bispectral index will be monitored
  Other Names: bispectral index monitor

SUMMARY:
Because neoplastic disease is one of the leading causes of death worldwide and breast cancer is one of the most frequent neoplasia among women, the possibility of influencing the evolution of patients starting from the moment of surgical intervention using a perianesthesic intervention is a scientific topic of high interest. The study will compare two anesthetic techniques and their efficiency in lowering the factors that can favorize the dissemination of neoplasia and their role in the prevention of postoperative pain. The serum level of vascular endothelial growth factor A (VEGF-A) will be determined before and after the surgical intervention after using two different types of anesthesia (inhalational and intravenous), and the immunohistochemical expression of vascular endothelial growth factor receptors (VEGFR) will be determined on the excised tissue. For the two different types of anesthesia a continuous infusion of lidocaine 1% will be associated. The study will compare the short-term and long term-outcome of the patients assigned the two different types of anesthesia and their immediate postoperative evolution .

DETAILED DESCRIPTION:
The study will enroll patients with ages between 18 and 80 years old, diagnosed with breast cancer but without proof of disease dissemination on medical imaging. After obtaining an informed consent the patients will be computer randomized to 4 groups. Each group will benefit from a certain type of anesthesia. The first group will be assigned general anesthesia using Sevoflurane for maintenance of hypnosis, the second group will be assigned general anesthesia with Sevoflurane and a continuous infusion of lidocaine 1%. The thrid group will be assigned total intravenous anesthesia using propofol for maintenance of hypnosis and the fourth group will be assigned to total intravenous anesthesia with propofol and a continuous infusion of lidocaine 1%. Before the surgical procedure a blood sample will be drawn from each patient for the measurement of serum vascular endothelial growth factor A ( VEGF-A). All the patients will receive pre-medication a night before the intervention with low molecular weight heparin (LMWH) and midazolam 5mg the morning of the intervention. For the first two groups the anesthetic induction will be conducted using propofol 1,5-2 mg/kg, fentanyl 1-3 microg/kg, atracurium 0,5 mg/kg.For the maintenance of anesthesia Sevoflurane will be used at a alveolar concentration of 1-1,5 MAC, as to maintain a BIS between 45-55. Intraoperative anesthesia will be ensured by using fentanyl boluses of 100 microg and the muscular relaxation needed for mechanical ventilation will be maintained using boluses of 10 mg of atracurium. At the end of the surgery the neuromuscular blockade will be antagonized with neostigmine 0.05 mg/kg and atropine 0.2 mg/kg. For the second group at the induction of anesthesia the patient will be administered a bolus of lidocaine 1% of 1.5 mg/kg and a continuous infusion of lidocaine 1% 2 mg/kg/h will be associated throughout the procedure and 1mg/kg/h,24 h postoperative. The postoperative analgesia will be assured by administering acetaminophen 1 g each 8 h and tramadol 25-50 mg each 4-6 h as needed. For the third and fourth groups the induction of aneshesia will be made using propofol administered by target controlled infusion (TCI) technique with a target plasma concentration of 4 microg/ml . Throughout the intervention the plasma concentration of propofol will be adjusted with increments of 0.2 microg/ml as to maintain a BIS between 45-55. To attenuate the response to laryngoscopy the patient will receive a bolus of fentanyl 1-3 microg/ml. During the intervention fentanyl will be administered in boluses of 100microg as needed. Muscular relaxation necessary for intubation will be provided using atracurium 0.5 mg/kg at induction of anesthesia and 10 mg boluses during the surgery as needed. At the end of the surgery the neuromuscular blockade will be antagonized with neostigmine 0.05 mg/kg and atropine 0.2 mg/kg. For the fourth group at the induction of anesthesia the patient will be administered a bolus of lidocaine 1% of 1.5 mg/kg and a continuous infusion of lidocaine 1% 2 mg/kg/h will be associated throughout the procedure and 1mg/kg/h, 24 h postoperative.Postoperative analgesia will be assured by administering acetaminophen 1 g each 8 h and tramadol 25-50 mg each 4-6 h as needed. Throughout the surgical intervention the patients will be monitored accordingly to the American Society of Anesthesiologists (ASA) standards (electrocardiogram-ECG, heart rate- HR, peripheral capillary oxygen saturation- SpO2, non-invasive blood pressure- NIBP, capnography and for the 3rd and 4th groups the bispectral index - BIS will be monitored). In the postoperative period non-invasive blood pressure -NIBP, heart rate- HR,peripheral capillary oxygen saturation SpO2, intensity of pain at 24 and 48 h will be monitored.Vascular endothelial growth factor- VEGF levels will be monitored at 24 h postoperative using ELISA technique. Vascular endothelial growth factor receptors 1 and 2 (VEGFR1 and VEGFR2) will be determined using immunohistochemical staining.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer
* ASA risk class I-III
* no metastatic disease

Exclusion Criteria:

* hepatic, pulmonary metastasis
* type I and II diabetes
* rheumatoid arthritis
* osteoarthritis
* ischemic cardiovascular disease (history of myocardial infarction, angina)
* peripheral vascular disease
* endometriosis
* allergies to lidocaine, fentanyl, propofol, sevoflurane, atracurium, midazolam, acetaminophen, tramadol
* neuropsychiatric disorders
* incapacity of understanding the study
* refusal of participation

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
serum concentration of vascular endothelial growth factor A (VEGF-A) | 1 year

SECONDARY OUTCOMES:
pain score | 1 year
  assesed using visual-analogue scale
survival of patients | up to 5 years
Vascular endothelial growth factor receptor 1 and 2 (VEGFR1 and VEGFR2) density | at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- IOCN Prof Dr I chiricuta, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mao L, Lin S, Lin J. The effects of anesthetics on tumor progression. Int J Physiol Pathophysiol Pharmacol. 2013;5(1):1-10. Epub 2013 Mar 8. PMID 23525301
- [Background] Byrne K, Levins KJ, Buggy DJ. Can anesthetic-analgesic technique during primary cancer surgery affect recurrence or metastasis? Can J Anaesth. 2016 Feb;63(2):184-92. doi: 10.1007/s12630-015-0523-8. PMID 26497721
- [Result] Chang YC, Liu CL, Chen MJ, Hsu YW, Chen SN, Lin CH, Chen CM, Yang FM, Hu MC. Local anesthetics induce apoptosis in human breast tumor cells. Anesth Analg. 2014 Jan;118(1):116-24. doi: 10.1213/ANE.0b013e3182a94479. PMID 24247230
- [Result] Terkawi AS, Sharma S, Durieux ME, Thammishetti S, Brenin D, Tiouririne M. Perioperative lidocaine infusion reduces the incidence of post-mastectomy chronic pain: a double-blind, placebo-controlled randomized trial. Pain Physician. 2015 Mar-Apr;18(2):E139-46. PMID 25794212
- [Derived] Galos EV, Tat TF, Popa R, Efrimescu CI, Finnerty D, Buggy DJ, Ionescu DC, Mihu CM. Neutrophil extracellular trapping and angiogenesis biomarkers after intravenous or inhalation anaesthesia with or without intravenous lidocaine for breast cancer surgery: a prospective, randomised trial. Br J Anaesth. 2020 Nov;125(5):712-721. doi: 10.1016/j.bja.2020.05.003. Epub 2020 Jun 29. PMID 32616309